CLINICAL TRIAL: NCT05736276
Title: Empathy Levels Among Undergraduate Medical Students in Karachi, Pakistan - a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Other Study IDs: 0110721MNY5
Record Dates: First submitted 2023-01-18; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Empathy
Keywords: empathy; medical students; Pakistan; surveys and questionnaires; observational study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Empathy is a concept native to the field of medicine. However, over the course of medical school, empathy levels are expected to decline. The aim of this study was to assess the empathy levels amongst medical students in relation to their year of study and specialties of choice in the future. A cross-sectional study was conducted to assess empathy levels among students from medical colleges in Karachi, Pakistan, using an online survey. The total duration of the study was two months. The authors analyzed the data using SPSS version 20. A total of 463 undergraduate medical students participated in this survey.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate medical students

Exclusion Criteria:

* all the remaining population

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Undergraduate medical students enrolled in different years of the academic program were involved to cater to those in the pre-clinical years as well as those receiving clinical exposure.
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Empathy score on the Jefferson Scale of Empathy (JSE) | June 2022 - July 2022
  The total score range of the JSE is 20-140. Each factor of the questionnaire attributes to both positive and negatively phrased questions with '1' signifying 'strongly disagree' and '7' signifying 'strongly agree'.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No